CLINICAL TRIAL: NCT06520059
Title: Comparison of Efficacy of Intraosseous vs Intra-articular Injections of PRP for Advanced Knee OA
Brief Title: Optimal Articular Solutions With Intraosseous and Synovial Platelet-Rich Plasma
Acronym: OASIS-PRP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, MD, MSC, MPH, PHD, FEBVS, Universidade do Porto
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-2024
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Injections, Intra-Articula;; Regenerative Medicine;; Cartilage Repair
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study is a prospective cohort, parallel design clinical trial comparing the efficacy of intraosseous versus intra-articular injections of PRP for treating advanced knee osteoarthritis. Patients are matched for sex and age, and outcomes are assessed using VAS scores, KOOS, and MRI evaluations over a 12-month period. The study aims to determine which injection method provides superior pain relief and functional improvement.
Who Masked: Investigator
Masking Description: In this study, blinding (masking) will be applied to the outcome assessors. Patients will notice which specific type of PRP injection (intraosseous or intra-articular) they are receiving. Outcome assessors who evaluate the VAS scores, KOOS, and MRI results will also be blinded to the group assignments to prevent bias in the assessment of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous and intra-articular PRP (Active Comparator): Two intraosseous injections of PRP and another intra-articular injection of PRP on the same day.
  Interventions: Combination Product: Platelet rich-plasma - PRP - intraosseous and intra-articular admnistration
- Intra-articular PRP (Active Comparator): Patients submited to two intra-articular injections of PRP, separated by one week.
  Interventions: Combination Product: Platelet rich-plasma - PRP - intraosseous and intra-articular admnistration

INTERVENTIONS:
Combination Product: Platelet rich-plasma - PRP - intraosseous and intra-articular admnistration — Group 1 will receive two intraosseous injections of PRP and a subsequent/synchronous intra-articular injection of PRP on the same day.
  Group 2 will only receive two intra-articular injections of PRP, separated by one week.

SUMMARY:
This is a prospective cohort clinical study. Due to logistic constraints at the sites of implementation, a randomized allocation will not be feasible (private clinic). Patients will be selected with the aim of matching for important confounders (sex and age) the grade of knee OA will be restricted to advance stages.

DETAILED DESCRIPTION:
A prospective cohort clinical study. The matched sample will be divided into two groups. Group 1 will receive two intraosseous injections of PRP and another intra-articular injection of PRP on the same day.

Group 2 will only receive two intra-articular injections of PRP, separated by one week. One week before the PRP injection, both groups will receive an intra-articular injection of 20 mg triamcinolone hexacetonide.

The PRP is obtained from an autologous blood sample. PRP production consists of a 54 mL (PRP intra-articular) and 80 mL (PRP intraosseous) sample of venous blood from the cubital vein of the patient's upper limb, using 6 x 9 ml tubes, containing a 3.2% sodium citrate solution. The tubes will be centrifuged at 2400 rpm for 12 minutes at room temperature. It is obtained a suspended concentration of PRP that is carefully extracted using a pipette to avoid aspiration of leukocytes from the buffy coat (leukocyte-poor PRP [LP-PRP]). For group 1, it will be injected 4 mL intraosseous, and 8 mL intra-articular. Group 2 will be injected 8 ml of PRP twice (one each week). A total of 8 ml of PRP will be injected into the knee.

A hemogram will be used to analyze the blood sample and the PRP to evaluate their characteristics (concentration of red blood cells, concentration of white blood cells, concentration of platelets, and mean platelet volume); with this analysis, it will be also calculated the platelet concentration growth factor (between baseline blood sample and PRP). Besides concentration, it will also be calculated the total volume of platelets injected into the knee.

All procedures will be carried out in a laminar flow chamber (0.34 m/s) to avoid contamination. Following preparation, the PRP will be injected with the minimum time elapsed since its preparation (maximum 30 minutes).

The PRP is injected after the skin is prepared and draped. If needed, synovial fluid aspiration will be done before injections. With the patient lying in a supine position on the examination table, with the knees fully extended, the PRP intra-articular injection is performed in a sterile manner via a superolateral patellar approach under ultrasound guidance (Logiq E R8, GE Healthcare).

Regarding intraosseous injections, the location and exploration of the joint line, tibial plateau, and femoral condyle will be done with ultrasound. Following the identification of the articular line through ultrasound examination, the two insertion points for the intraosseous infiltrations in the knee are marked: 2 cm below the tibiofemoral joint line for the tibial plateau and 2 cm above the tibiofemoral joint line for the femoral condyle. The procedure is done for the affected knee compartment (medial or lateral).

To ensure effective and safe analgesia during the intraosseous infiltration procedure, a solution of 1% lidocaine (10 mg/mL). In summary, a 10 mL syringe will be filled with the previously mentioned specified solution and then injected at the marked points-the tibial plateau and femoral condyle. Approximately 4-5 mL will be injected along the path until contact is made with the periosteum, where the trocar will be inserted. An additional 4-5 mL will be injected after the insertion of the trocar. A 10-20 minute time interval will be observed before proceeding with the intraosseous infiltrations. The tibial plateau and femoral condyle will be targeted, and a 15-G trocar-biopsy needle system (1.8 mm diameter, 90 mm length, Arrow OnControl Aspiration needle set, Teleflex Medical Europe Ltd., Dublin, Ireland) will be placed on the tibial and condyle entry mark points. Subsequently, the trocar will be attached to a power driver (Arrow OnControl Powered Bone Access System, Teleflex Medical Europe Ltd., Dublin, Ireland) encased in a sterile plastic sleeve. The trocar will be advanced with precision while its placement is verified using ultrasound imaging. It will be positioned 2 cm below the articular line at a 45-degree angle in the tibial plateau, and 2 cm above the articular line at a 30-degree angle, penetrating 1.5-2 cm into the bone. Accurate depth measurement is made with laser marks on the trocar, spaced 1 cm apart. Once the correct position is confirmed, the power driver will be detached, and the needle core removed. Afterward, 6 mL of activated PRP will be injected through the trocar. Following the injection, the needle core will be reinserted and reattached to the power driver, and the trocar will be withdrawn. Intraosseous infiltration will be consistently performed at the same site in all procedures, as PRP is expected to distribute uniformly across the subchondral area regardless of tissue lesions.

After injection, patients are allowed to mobilize the knee joint, walk as desired and are instructed to apply ice over the injected area for the next 24-48 hours. Patients will be requested to avoid vigorous activity for a minimum of 10 days and to avoid taking NSAIDs for 7 days after injection. Consumption of acetaminophen (max 3 gm/day) will be allowed in the management of pain during the post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals with unilateral or bilateral symptomatic knee OA diagnosis according to the American College of Rheumatology
* with symptoms for more than 3 months
* confirmed with radiologic diagnosis (Kellgren-Lawrence grades III or IV).
* Patients must be able to walk with a painful knee.

Exclusion Criteria:

* previous history of knee surgery
* systemic autoimmune or rheumatic disease
* platelet diseases
* use of NSAIDs 3 days prior the injections
* previous history (last 3 months) of systematic use of corticosteroids
* or other intra-articular injections in the knee in the past 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PROM - Knee related Qol | baseline, and at follow-up of 3 months, 6 months and 12 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) - absolute value from the score (units). Min-Max (0-100) higher scores indicate better outcomes and a higher quality of life related to the knee
PROM - PAIN | baseline, and at follow-up of 3 months, 6 months and 12 months
  Visual analogic Score - PAIN (VAS) -absolute value from the score (units). Min-Max (0-10) higher scores indicate worse outcomes

SECONDARY OUTCOMES:
bone marrow edema -MRI | 1 month prior to the injection; 1 month to one year after intervention
  first scored dichotomous (yes/no)
bone marrow edema -MRI | 1 month prior to the injection; 1 month to one year after intervention
  BME will be classified using the criteria defined in the Whole-Organ Magnetic Resonance Imaging Score (WORMS). Range 0-3 Higher scores mean more medular edema.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
This experimental study is safe for patients and will be carried out according to the principles of the Declaration of Helsinki and the European Union General Data Protection Regulation (GDPR). All data processing will be anonymous.